CLINICAL TRIAL: NCT02681835
Title: Comparison of the C-MAC and Macintosh Laryngoscopes for Tracheal Intubation in Different Intubator Positions. A Randomized, Crossover, Manikin Trial
Brief Title: Endotracheal Intubation in Prehospital Scenario
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02.007.1MR
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Endotracheal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Position 1 (Experimental): Standard position during intubation. Intubator is behind head of the victim, propped up on both elbows
  Interventions: Device: C-MAC laryngoscope; Device: Macintosh laryngoscope
- Position 2 (Experimental): Intubator is behind head of the victim, lies on the left side
  Interventions: Device: C-MAC laryngoscope; Device: Macintosh laryngoscope
- Position 3 (Experimental): Intubator stands astride the victims, intubated using the face-to-face
  Interventions: Device: C-MAC laryngoscope; Device: Macintosh laryngoscope

INTERVENTIONS:
Device: C-MAC laryngoscope — Intubation performed using C-MAC laryngoscope
  Other Names: C-MAC
Device: Macintosh laryngoscope — Intubation performed using laryngoscope with Macintosh blade
  Other Names: C-MAC

SUMMARY:
We therefore designed this randomized crossover study to compare C-MAC with Macintosh laryngoscope in emergency intubation performed by paramedics according to three different intubator positions.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* maximum 1 year of work experience in medicine
* minimum 50 clinical intubations
* paramedics

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time required for successful intubation | 1 day

SECONDARY OUTCOMES:
success rate of intubation attempt | 1 day
  success rate of first, second and third intubation attempt
cumulative success ratios related to time | 1 day
  cumulative success ratio was counted as percentage of successful intubations in time intervals in all scenarios
Ease of intubation | 1 day
  To access subjective opinion about the difficulty of each intubation method, participants were asked to rate it on a visual analog scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).
Cormack&Lehane grade | 1 day
  glottic view during intubation rate using Cormack&Lehane grade
Dental Compression | 1 day
  the severity of the potential dental trauma was calculated based on previously described modified grading scale (Svoldelli, 2009)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided